CLINICAL TRIAL: NCT06863727
Title: The Beijing Longitudinal Disability Survey in Community Elderly
Acronym: BLINDSCE
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Sponsor
Other Study IDs: No.[2023]129; 2024-2G-20112 (Other Grant/Funding Number: Capital's Funds for Health Improvement and Research)
Record Dates: First submitted 2025-02-16; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ageing; Disability; Cognitive Impairment; Frailty; Intrinsic Capacity
Keywords: Ageing; Disability; Cognitive Impairment; Community; Cohort
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plan to obtain blood samples from some of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to establish the prospective cohort of the Beijing Longitudinal Disability Survey in Community Elderly (BLINDSCE) to explore the high-risk factors and preventive interventions for disability and cognitive impairment among community-dwelling adults aged 65 years and over. The main question it aims to answer is:

* What are the high-risk factors able to predict the incidence and advance of disability and cognitive impairment in community-dwelling adults aged 65 years and over?
* What are the categories of function and cognitive performance trajectory in community-dwelling adults aged 65 years and over?

DETAILED DESCRIPTION:
BLINDSCE is a community-based prospective cohort study that includes individuals aged 65 and over from urban and rural areas in Beijing. Participants will provide detailed demographic information and undergo multifactorial questionnaires, disability measurements, cognitive assessments, other disability-related outcomes, and clinical biochemical measures. The study has started recruitment and enrollment in 2023 and will follow-up once every 1-2 year. This work consists of three steps as follows. First, by collecting baseline and follow-up data of participants, we plan to establish a community-dwelling elderly database in Beijing. Second, high-risk factors can be pre-screening based on this cross-sectional analysis. Third, longitudinal data was used to develop the prediction model and trajectory analysis for disability and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged 65 years or older who reside in Beijing.
* Participants who sign an institutionally approved informed consent.

Exclusion Criteria:

* Participants with severe mental disorders and serious medical conditions preventing study investigation
* Participants undergoing long-term professional treatment for physical function and cognitive functioning, such as hospitalization or rehabilitation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community residents aged 65 years or older in Beijing
Sampling Method: Non-Probability Sample
Enrollment: 1962 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Disability from the individual's perspective | An average of 1 to 2 years
  Disability is assessed using the 12-item World Health Organization's Disability Assessment Schedule 2.0 (WHODAS 2.0). The WHODAS 2.0 is a patient-reported disability measure, comprising six life domains involving cognition, mobility, self-care, interpersonal relationships, life activities, and participation. The total score of 12-item WHODAS 2.0 categorizes disability from no disability (score 0) to complete disability (score 48).
Disability from the medical's perspective | An average of 1 to 2 years
  Disability is assessed using the basic activities of daily living (BADL) scale, the Katz Index scale. The minimum value is 0 , and the maximum value is 6. The higher the score, the better the outcome.
Disability from the medical's perspective | An average of 1 to 2 years
  Disability is assessed using the instrumental activities of daily living (IADL) scale, the Lawton and Brody IADL scale. The minimum value is 0, and the maximum value is 8. The higher the score, the better the outcome.

SECONDARY OUTCOMES:
Cognitive impairment | An average of 1 to 2 years
  The cognitive impairment is assessed by the Mini-Mental State Examination (MMSE). The minimum value is 0, and the maximum value is 30. The higher the score, the better the outcome.
Cognitive impairment | An average of 1 to 2 years
  The cognitive impairment is assessed by the Montreal Cognitive Assessment-Basic (MoCA-B). The minimum value is 0, and the maximum value is 30. The higher the score, the better the outcome.
Subjective cognitive decline | An average of 1 to 2 years
  Subjective cognitive decline is assessed by the subjective cognitive decline questionnaire-9 items (SCD9). The minimum value of SCD9 is 0, and the maximum value is 9, the higher the score, the worse the outcome.
Intrinsic capacity | An average of 1 to 2 years
  Intrinsic capacity is the composite of physical and mental abilities that an individual can draw upon. It comprises locomotor, sensory (hearing and vision), vitality, psychological, and cognition domains. The intrinsic capacity composite score is used to assess intrinsic capacity. The intrinsic capacity composite score ranges from 0 to 100, and the higher the score, the better the outcome.
Intrinsic capacity | An average of 1 to 2 years
  Intrinsic capacity is assessed by the integrated care for older people (ICOPE) scale. The minimum value of the ICOPE score is 0, and the maximum value is 5, the higher the score, the better the outcome.
Frailty | An average of 1 to 2 years
  Frailty is assessed using the Fried frailty phenotype (FFP) scale. The minimum value is 0, and the maximum value is 5. The higher the score, the worse the outcome.
Hospitalization | An average of 1 to 2 years
  Hospitalized times, duration, diagnosis, surgery, bedridden status, assisted ventilation treatment, catheter treatment are collected by questionnaire and supplemented through a review of electronic medical records.
Death | An average of 1 to 2 years
  The date and cause of death are collected from the participant's family members/healthcare providers and supplemented through a review of electronic medical records.
Appendicular skeletal muscle mass | An average of 1 to 2 years
  Appendicular skeletal muscle mass (ASM) is estimated using a physical measurement formula. Weight in kilograms, height in centimeters, gender(male or female), and age in years are combined to report ASM through the formula: ASM = 0.193*weight(kg) + 0.107*height(cm) - 4.157 * gender - 0.037*age(year) - 2.631. The higher the value, the better the outcome.
Muscle strength | An average of 1 to 2 years
  Muscle strength is assessed by the grip strength. The higher the value, the better the outcome.
Physical performance | An average of 1 to 2 years
  Physical performance is assessed by the Short Physical Performance Battery (SPPB) test. The minimum score is 0, and the maximum score is 12. The higher the score, the better the outcome.
Sarcopenia | An average of 1 to 2 years
  Sarcopenia is screened by the SARC-F scale. The minimum value is 0, and the maximum value is 10. The higher the score, the worse the outcome.
Sarcopenia | An average of 1 to 2 years
  Sarcopenia is assessed based on the criteria recommended by the Asian Working Group for Sarcopenia (AWGS) 2019 consensus, including muscle strength, plus appendicular skeletal muscle mass (ASM), and/or physical performance. AWGS 2019 contends that diagnosing sarcopenia requires both low muscle strength and muscle mass, and defines persons with low muscle mass, low muscle strength, and low physical performance as having "severe sarcopenia."

CONTACTS AND LOCATIONS:
Overall Officials: Yansu Guo, Ph.D, Principal Investigator — Beijing Geriatric Healthcare and Disease Prevention Center, Xuanwu Hospital, Capital Medical University
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cheng S, Du X, Hou C, Liu H, Lei S, Wu Y, Yue X, Guo Y. Beijing Longitudinal Disability Survey in Community Elderly (BLINDSCE): protocol for a community-based prospective longitudinal cohort study about disability prediction model. BMJ Open. 2025 May 15;15(5):e091955. doi: 10.1136/bmjopen-2024-091955. PMID 40379348